CLINICAL TRIAL: NCT03572036
Title: Long-term Clinical Outcomes of Phosphodiesterase Type-5 Inhibitor Therapy in Sickle Cell Patients With Pulmonary Hypertension
Brief Title: Phosphodiesterase Type-5 Inhibitor Therapy in Sickle Cell People With Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999918109; 18-H-N109
Record Dates: First submitted 2018-06-27; First posted 2018-06-28 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Hypertension; Sickle Cell Disease
Keywords: Outcomes Assessment; Sickle Cell Disease
MeSH Terms: conditions — Hypertension, Pulmonary; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arm 1: aged 18 and older, participated in 001-H-0088 and 04-H-0161 and 1) a diagnosis of SCD 2) a diagnosis of PH 3) prescribed and/ or reported taking PDE5-I therapy for a duration of >16 weeks.

SUMMARY:
Background:

Sickle cell disease (SCD) is a common inherited blood disorder. Many people with SCD are at risk to get pulmonary hypertension (PH). PH means that the blood pressure in the blood vessels to the lungs is high, and is a serious disease and. Very few studies have looked at the success of treatments for PH in people with SCD. Researchers want to learn more about treating PH with a type of drug called phosphodiesterase type 5 inhibitors (PDE5-I). They will look at the records of people who have already joined other studies.

Objective:

To identify people who already joined NIH SCD protocols whose medical records should be reviewed. The review will look at the description of SCD patients with PH who have already taken PDE5-I and the outcomes for these people.

Eligibility:

Adults ages 18 and older with SCD and PH. They must have joined certain NIH studies and taken PDE5-I therapy for at least 16 weeks.

Design:

This study is a review of medical records.

Researchers will collect data from databases of existing studies. They will identify people in those studies who have SCD and PH and took the study drug for at least 16 weeks.

Researchers will review the full medical records of those people.

From that review, researchers will find participants who meet the inclusion criteria. They will extract data from those records.

Researchers will analyze the data. This includes results from heart and lung tests, imaging, and walking tests. It will also include results of a procedure called right heart catheterization.

Demographic data and lab data will also be collected.

Researchers will remove identifying information from the data, then share it in a database.

DETAILED DESCRIPTION:
There is a lack of evidence-based treatment for patients with sickle cell disease (SCD) with pulmonary hypertension (PH). PH is a leading cause of mortality in SCD and is an independent risk factor for mortality in this population. SCD is a major health problem worldwide, primarily affecting people of African descent. In the United States approximately 100,000 individuals have SCD and 0.2% of African Americans have homozygous SS sickle cell disease, while 8% of African Americans carry one allele and have sickle cell trait. In developed countries, even in the current era of hydroxyurea, SCD patients have relatively shortened lifespans with a median life expectancy of approximately 48 years for females and 42 years for males.

PH affects up to 1/3 of adults screened by echocardiography and pre-capillary PH is diagnosed in 6% by right heart catheterization (RHC). Data suggest that either precapillary or post-capillary PH in SCD are associated with a 5-fold risk of early mortality, and SCD subjects with echocardiographic signs of both have a 13-fold risk of early mortality. Though a cause and effect relationship between the presence of PH and early mortality in adult subjects with SCD has not been conclusively established, data regarding the causes of death in a prospective observational study of adult SCD patients suggest that cardiopulmonary cause of death was present in at least 35% of patients.

The World Health Organization (WHO) reclassified SCD-related PH as Group 5 in 2013. Therefore, SCD-related PH is not eligible for vasodilator therapies currently available for WHO Group 1 pulmonary arterial hypertension (PAH). There have only been three prospective clinical trials of vasodilator therapies in sickle cell patients with RHC-defined PH. After the findings of the Walk-PHaSST study were reported, a strong recommendation against sildenafil in sickle cell patients with PH was made in guidelines published by the American Thoracic Society in 2014. However, a major limitation of the trial was that, in order to improve trial feasibility, subjects were eligible for enrollment based on an elevated TRV, as well as RHC-defined PH, leading to incomplete hemodynamic characterization of study patients. The physiologic understanding of the differences between subjects who developed SAEs and those who tolerated sildenafil remains poorly understood. In individual circumstances, some patients may have chosen to continue sildenafil. If some patients with SCD-related PH have continued to benefit from sildenafil therapy in the time since this clinical trial was reported, it would raise the question of whether a subgroup of SCD-related PH patients may still benefit from PDE5-Is and how these patients could be clinically characterized.

Given the difficulty of enrolling SCD-related PH patients into prospective, multi-center trials, for example as demonstrated by the ASSET trials being closed due to low enrollment, we plan to utilize existing clinical data available on patients who were documented to have RHC- defined PH prior to initiation of PDEI-5 therapy, in order to better characterize the use of this medication in patients with SCD-related PH.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects aged 18 and older, participated in 001-H-0088 and 04-H-0161
* a diagnosis of SCD
* a diagnosis of PH by right heart catheterization
* prescribed and/ or reported taking PDE5-I therapy for a duration of greater than or equal to 16 weeks. (We will not be able to use medication dispensation records alone to verify whether subjects were compliant as not all medications were dispensed directly from the NIH pharmacy.)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects aged 18 and older, participated in 001-H-0088 and 04-H-0161 and 1) a diagnosis of SCD 2) a diagnosis of PH 3) prescribed and/ or reported taking PDE5-I therapy for a duration of >16 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Perform multivariable regression analyses for factors associated with morbidity and mortality | At the end of data analysis
  We hypothesize that there are some subjects, for example those with RHC-defined PH, with particular characteristics who may benefit from improved morbidity and mortality with the use of long- term PDE5-I therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Swee Lay Thein, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States